CLINICAL TRIAL: NCT06577662
Title: Effects of an Individual and Family Self-Management of Fall Prevention Program on Balance Ability and Fall-related Self-efficacy Among Chinese Post-Stroke Individuals
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chiang Mai University (Other)
Collaborators: The Affiliated Hospital Of Guizhou Medical University (Other)
Responsible Party: Principal Investigator, Wang Yinhua, Head nurse, Chiang Mai University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2567-FULL018
Record Dates: First submitted 2024-08-27; First posted 2024-08-29 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Stroke, Ischemic; Self Efficacy; Fall
MeSH Terms: conditions — Ischemic Stroke | interventions — Laboratory Proficiency Testing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- individual and family self-management (IFSM) fall prevention program (Experimental): The IFSM program will be last for ten weeks, two weeks in the hospital, and follow up at eight weeks after patients discharge to home. It includes 11 sessions, including ten sessions developed in the inpatient department within two weeks and one online booster session developed in the first month (week 4) after discharge in home. There will be also one session just for caregivers, which aims to improve caregivers' skills to keep patients' safety. In the process, self-efficacy strategies, self-regulation skills, and social facilitation are used in every session. The main self-efficacy strategies includes skill mastery, vicarious experience, and verbal persuasion. Several self-regulation skills for patients and caregivers are also used in the study, such as self-monitoring and reflective thinking. A WeChat group will be established to support patients and their families.
  Interventions: Behavioral: individual and family self-management (IFSM) fall prevention program
- usual care (No Intervention): Participants in the control group will receive usual care, including standard clinical practices such as education on fall prevention and a fall prevention booklet. The education will be delivered by the researcher and does not include any additional intervention specific to the study. A fall prevention care plan will be manually documented in the electronic health record. After the patients are discharged home, a phone visit will be provided for patients within the first month, which will include a medication review and professional access. Participants will also use a fall record diary to record falls in the control group, and this will be copied for data extraction after the experiment.

INTERVENTIONS:
Behavioral: individual and family self-management (IFSM) fall prevention program — The IFSM program will last for ten weeks, two weeks in the hospital, and follow up at eight weeks after patients discharge to home. It will include 11 sessions, including ten sessions developed in the inpatient department within two weeks and one online booster session developed in the first month (week 4) after discharge in home. There will be also one session just for caregivers.
  Session 1 : PRST combined with GRI (one) Session 2 : Environment safety Session 3 : Assistant technology Session 4 : PRST combined with GRI (two) Session 5 : Medication review Session 6 : Safety in daily activities Session 7 : How to keep loved one safety Session 8 : Review of PRST combined with GRI Session 9 : Review of other five fall prevention skills Session 10 : Summary of the program and setting goals Session 11 : Booster session Week 10: Evaluation
  Arms: individual and family self-management (IFSM) fall prevention program

SUMMARY:
This study is about exploring the effectiveness of individual and family self-management (IFSM) fall prevention programs on balance ability and fall-related self-efficacy in post-stroke people. The main intervention measures were developed based on the risk and protective factors of fall prevention in post-stroke people, including exercise, environment safety, assistant technology, medication review, and safety in daily activities. The intervention was implemented in 10 weeks for both patients and their family members. By mastering these skills, post-stroke people may reduce the number of falls after discharge to home.

ELIGIBILITY:
Inclusion Criteria:

* For patients

  * aged 18 years or above;
  * first-ever diagnosed with ischemic stroke;
  * level of impairment assessed by the National Institutes of Health Stroke Scale (NIHSS) scores between 5 to 15 (moderate severity) before entering the experiment;
  * mental state assessed by Mini-Mental State Exam score > 24;
  * mobility tested by Timed Up and Go ≥12.6 second (walkers or another kinds of gait aid are allowed to be used in the test);
  * motor power of all limbs examined by muscle power assessment grade ≥3;
  * ability to understand Chinese;
  * living with family members;
  * having phones that can use the internet;
  * willing to join the study.
* For caregivers

  * mental state assessed by Short Portable Mental Status Questionnaire score ≥8;
  * being the primary caregiver, living in the same house, and taking care of the patient;
  * having phones that can use the internet;
  * can speak, understand, and write in Chinese; and (e) willing to participate.

Exclusion Criteria for patients:

* having problems with sensory and/or global aphasia

Discontinuation criteria:

* patients have an illness that needs hospitalization;
* patients and caregivers cannot complete participation in intervention sessions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Fall-related self-efficacy | Fall-related self-efficacy will be measured before the fall prevention program and after patients are discharged in 8 weeks.
  Fall-related self-efficacy refers to the level of perceived confidence in undertaking everyday activities without falling, which includes self-efficacy in balance ability, preventing falls, and managing falls. The Short Falls Efficacy Scale-International (Short FES-I) will be used to assess fall-related self-efficacy; it consists of seven questions. A four-point scale is used to score each item, and a higher score indicates lower self-efficacy. The total score is calculated by adding the scores of each item, giving a scale ranging from 7 to 28 for the seven items. The Short FES-I has previously demonstrated excellent reliability (Cronbach's α = 0.92).
Balance ability | Balance ability will be measured before the fall prevention program and after patients are discharged in 8 weeks.
  Balance ability is the ability to maintain the body's stability, including keeping a certain posture or balance when subjected to external forces. Berg Balance Scale (BBS) will be used to assess the balance ability in post-stroke people. The BBS will be used to assess balance ability in post-stroke individuals. It consists of 14 items, each rated on a five-point scale. A score of 41-56 indicates the ability to walk independently, 21-40 indicates the ability to walk with assistance, and 0-20 indicates wheelchair-bound movement. In different studies on patients with stroke, the BBS has been found to have excellent internal consistency, with Cronbach alphas ranging from 0.92 to 0.98

SECONDARY OUTCOMES:
Number of falls, fall-related injuries and Adverse Events | Number of falls and fall-related injuries will be measured after patients are discharged in 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated hospital of Guizhou Medical University, Guiyang, Guizhou, China

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant-level data related to the primary and secondary outcomes
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Individual participant data (de-identified) will be available upon reasonable request from the corresponding author. The data will be available beginning 6 months after publication for a period of 3 years. Data will be shared for academic purposes only.
Access Criteria: Access to the de-identified individual participant data (IPD) and supporting documentation (such as the study protocol, statistical analysis plan, and informed consent form) will be granted to qualified researchers affiliated with academic or non-profit institutions.
  Researchers must submit a methodologically sound research proposal along with a data access request to the corresponding author. The request will be reviewed by the study team to ensure alignment with the original study objectives and participant privacy protections.
  Upon approval, a data use agreement will be signed. Data will be shared via secure email or a secure file-sharing platform, depending on the nature and size of the data.

REFERENCES:
- [Derived] Wang Y, Chaiard J, Lirtmunlikaporn S, Suwankruhasn N. Effects of an individual and family self-management of fall prevention programme on balance ability and fall-related self-efficacy among Chinese poststroke individuals: a study protocol for a randomised controlled trial. BMJ Open. 2025 Jul 15;15(7):e100966. doi: 10.1136/bmjopen-2025-100966. PMID 40664404